CLINICAL TRIAL: NCT05061381
Title: Evaluating the Impact of a School Wellbeing Programme on Internalising Problems in Primary School Children
Brief Title: Effectiveness of a School Wellbeing Programme for Internalising Problems in Irish Primary School Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University College Dublin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: aclancy
Record Dates: First submitted 2021-09-07; First posted 2021-09-29 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-07

CONDITIONS: Anxiety; Low Mood
MeSH Terms: conditions — Anxiety Disorders; Consciousness Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A Lust for Life Schools Programme Group (Experimental): A Lust for Life programme will be delivered to primary school pupils by their school teachers in six weekly lessons. Well-being and resilience will be promoted in each lesson through classroom discussions, videos, classroom activities and homework assignments.
  Interventions: Behavioral: A Lust for Life Schools Programme
- Waiting list control group (No Intervention): Participants will be placed on a sixteen-week waiting list for the programme.

INTERVENTIONS:
Behavioral: A Lust for Life Schools Programme — A Lust for Life is a universal school-based multi-component programme whose target is to build well-being and emotional resilience in children. The programme was informed by evidence-based psychological approaches including mindfulness, cognitive behaviour therapy and positive psychology. It is delivered in six weekly lessons by the childrens' school teacher and involves classroom discussions, videos, classroom activities and homework assignments.
  Arms: A Lust for Life Schools Programme Group

SUMMARY:
The aim of this study is to assess the effectiveness of a school-based multi-component universal programme for the reduction of internalising problems (i.e. anxiety and low mood) in primary school pupils.

DETAILED DESCRIPTION:
Childhood and adolescence are important developmental phases for wellbeing and mental health. School has been noted in psychological literature to be a favourable environment for mental health initiatives, such as school-based programmes. Universal programmes are programmes delivered to all pupils irrespective of perceived need and have several advantages, including having a wide reach, avoiding the need for screening and are less stigmatising.

A Lust for Life is a universal school-based multi-component intervention whose target is to build well-being and emotional resilience in children. The programme was informed by evidence-based psychological approaches including cognitive behaviour therapy, positive psychology and mindfulness and consists of six lessons, each delivered by the pupils' school teacher on a weekly basis. The lessons involve classroom discussions, videos, classroom activities and homework assignments.

Study participants will complete the Revised Children's Anxiety and Depression Scale Short Format, Coping strategy indicator and Self-Efficacy Questionnaire for Children pre-intervention. Following this, schools randomly assigned to the experimental group will receive A Lust for Life, while those randomly assigned to the control group will be placed on a sixteen-week waiting list. The questionnaire measures and a Brief Satisfaction Scale will be completed by participants at post-intervention. In addition, a six-week follow-up assessment will determine whether the effects of the programme are sustained over a period of time. The programme will be delivered in the waiting list control group schools after the six-week follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

* Child
* Enrolled in primary school in Ireland
* Obtain written informed consent from parents/guardians
* Provide written assent

Exclusion Criteria:

* Failure to meet inclusion criteria

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 400 (Actual)
Dates: Start 2021-10-11 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-11-30 (Estimated)

PRIMARY OUTCOMES:
Symptoms of anxiety and low mood measured by the Revised Children's Anxiety and Depression Scale Short Form | 16 weeks
  25-item self-report measure of anxiety and depression symptoms of individuals aged 8-18 years.

SECONDARY OUTCOMES:
Coping skills as measured by the Coping Strategy Indicator | 16 weeks
  33-item measure that measures three coping factors: seeking social support, problem-solving, and avoidance.
Self-efficacy as measured by the Self-Efficacy Questionnaire for Children | 16 weeks
  24-item questionnaire that measures three factors: academic, social and emotional self-efficacy.

OTHER OUTCOMES:
Satisfaction with the programme measured by the Brief Satisfaction Scale | 10 weeks
  Scores on each item of the Brief Satisfaction Scale range from 1 to 7

CONTACTS AND LOCATIONS:
Overall Officials: Aoife Clancy, Principal Investigator — University College Dublin
Locations (1):
- University College Dublin, Dublin, Tipperary, Ireland

IPD SHARING:
Plan to Share IPD: Yes
The de-identified data collected in this research will be archived. Other researchers may contact the investigators to access the de-identified data for use in research into anxiety, depression, coping skills and self-efficacy.
Time Frame: The data collected in this study will be made available for other researchers after a manuscript reporting on the study's findings has been accepted for publication.
Access Criteria: Data may be accessed for use in research into anxiety, depression, coping skills and self-efficacy.